CLINICAL TRIAL: NCT00987337
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study To Evaluate The Safety And Efficacy Of Filibuvir Plus Pegylated Interferon Alfa-2a And Ribavirin In Treatment-Naive, HCV Genotype 1 Infected Subjects
Brief Title: Filibuvir In Treatment Naive Hepatitis C Virus (HCV) Genotype 1 Subjects
Acronym: FITNESS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A8121014
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Results first posted 2014-01-27 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2013-12

CONDITIONS: Hepatitis; Hepatitis C
Keywords: Hepatitis C Polymerase Inhibitor PF-00868554 Filibuvir
MeSH Terms: conditions — Hepatitis; Hepatitis C | interventions — filibuvir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A (Experimental): Filibuvir 300 mg BID + pegIFN/RBV x 24 weeks (subjects with undetectable HCV RNA at week 4)
  - or - Filibuvir 300 mg BID + pegIFN/RBV x 24 weeks followed by pegIFN/RBV x 24 weeks (subjects with detectable HCV RNA at week 4)
  Interventions: Drug: Filibuvir
- Arm B (Experimental): Filibuvir 600 mg BID + pegIFN/RBV x 24 weeks (subjects with undetectable HCV RNA at week 4)
  - or - Filibuvir 600 mg BID + pegIFN/RBV x 24 weeks followed by pegIFN/RBV x 24 weeks (subjects with detectable HCV RNA at week 4)
  Interventions: Drug: Filibuvir
- Arm C (Placebo Comparator): Placebo + pegIFN/RBV x 24 weeks followed by pegIFN/RBV x 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Filibuvir — 300 mg BID
  Arms: Arm A
Drug: Filibuvir — 600 mg BID
  Arms: Arm B
Drug: Placebo — BID
  Arms: Arm C

SUMMARY:
The primary objective for this study is to determine if the addition of filibuvir to a standard regimen of peginterferon/ribavirin (pegIFN/RBV) significantly increases the proportion of subjects who achieve a sustained viral response (SVR) compared to peginterferon/ribavirin (pegIFN/RBV) therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects at least 18 years of age.
* HCV seropositive.
* HCV RNA >10,000 IU/mL at screening.
* HCV Genotype 1. Subjects infected with a non-genotype 1 strain or mixed genotypes are not eligible.
* Treatment naïve (no prior treatment with IFN alfa +/ RBV regimens or investigational anti-HCV agents).
* Liver biopsy within two years (24 months) of Screening with non-cirrhotic fibrosis classification. For those subjects with liver biopsy outside of the time window or for those subjects with no history of liver biopsy, a biopsy must be performed prior to randomization.
* Ultrasound within 6 months of Screening for 1) those subjects with bridging fibrosis or 2) those subjects with AFP >50 and <100 ng/mL with no evidence of hepatocellular carcinoma. For those subjects with an ultrasound conducted outside the 6-month time window, an ultrasound must be performed prior to randomization.

Exclusion Criteria:

* Co-infection with either HIV or HBV.
* Evidence of severe or decompensated liver disease.
* Subjects with liver disease unrelated to HCV infection.
* Pre-existing medical condition that makes the subject unsuitable for treatment with pegIFN/RBV therapy per product labeling.
* Laboratory abnormality at Screening that makes the subject unsuitable for treatment with pegIFN/RBV therapy per product labeling.
* Abnormal ECG suggestive of clinically significant cardiac disease or QTc>450msec.
* History of organ transplant.
* Contraindicated medications being taken by the subject at the time of randomization that must be continued during the study period, including potent CYP3A4 inhibitors, sensitive CYP3A4 substrates, CYP3A4 substrates with narrow therapeutic range and CYP3A4 inducers.
* Active alcohol or substance abuse sufficient, in the Investigator's judgment, to prevent adherence to study medication and/or follow up.
* Pregnant or nursing females.
* Males whose female partner is pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2009-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (59):
- United States (25):
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, Coronado, California
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, Mather, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Englewood, Colorado
  - Pfizer Investigational Site, DeLand, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, South Miami, Florida
  - Pfizer Investigational Site, Winter Park, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Richmond, Virginia
- Belgium (5):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Edegem
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Haine-Saint-Paul
  - Pfizer Investigational Site, Leuven
- Canada (4):
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, Montreal, Quebec
- France (7):
  - Pfizer Investigational Site, Clichy
  - Pfizer Investigational Site, Créteil
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Pessac
  - Pfizer Investigational Site, Rennes
  - Pfizer Investigational Site, Vandœuvre-lès-Nancy
- Germany (6):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Bonn
  - Pfizer Investigational Site, Cologne
  - Pfizer Investigational Site, Düsseldorf
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Kiel
- Hungary (5):
  - Pfizer Investigational Site, Békéscsaba
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Debrecen
  - Pfizer Investigational Site, Gyula
  - Pfizer Investigational Site, Kaposvár
- Pfizer Investigational Site, Rio Piedras, Puerto Rico
- Pfizer Investigational Site, Seoul, South Korea
- Spain (5):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Córdoba, Cordoba
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Majadahonda, Madrid
  - Pfizer Investigational Site, Seville, Sevilla

REFERENCES:
- [Derived] Rodriguez-Torres M, Yoshida EM, Marcellin P, Srinivasan S, Purohit VS, Wang C, Hammond JL. A phase 2 study of filibuvir in combination with pegylated IFN alfa and ribavirin for chronic HCV. Ann Hepatol. 2014 Jul-Aug;13(4):364-75. PMID 24927607
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8121014&StudyName=Filibuvir%20In%20Treatment%20Naive%20Hepatitis%20C%20Virus%20%28HCV%29%20Genotype%201%20Subjects

RESULTS

PARTICIPANT FLOW:
Groups:
- Filibuvir 300 mg Plus pegIFN/RBV: Filibuvir 300 milligram (mg) tablet orally twice daily as blinded therapy along with pegylated interferon alpha-2a (pegIFN alpha-2a) 180 microgram (mcg) subcutaneously once weekly and ribavirin (RBV) 1000 milligram per day (mg/day) to participants weighing less than or equal to(<=) 75 kilogram (kg) or RBV 1200 mg/day to participants weighing greater than (>) 75 kg, orally in 2 divided doses up to Week 24. Participants with undetectable hepatitis C virus (HCV) ribonucleic acid (RNA) (HCV RNA <15 international units/milliliter [IU/mL]) from Week 4 through 24 were discontinued from therapy and followed through Week 72. Participants with detectable HCV RNA (greater than or equal to [>=] 15 IU/mL) at Week 4 or later but undetectable at Week 24 received open-label pegIFN alpha-2a 180 mcg subcutaneously once weekly and RBV 1000 mg/day if participant weighed <=75kg or RBV 1200 mg/day if participant weighed >75 kg, orally in 2 divided doses up to Week 48 and then followed through Week 72.
- Filibuvir 600 mg Plus pegIFN/RBV: Filibuvir 600 mg tablet orally twice daily as blinded therapy along with pegIFN alpha-2a 180 mcg subcutaneously once weekly and RBV 1000 mg/day to participants weighing <=75 kg or RBV 1200 mg/day to participants weighing >75 kg orally in 2 divided doses up to Week 24. Participants with undetectable HCV RNA (plasma HCV RNA <15 IU/mL) from Week 4 through 24 were discontinued from therapy and followed through Week 72. Participants with detectable HCV RNA (>=15 IU/mL) at Week 4 or later but undetectable at Week 24 received open-label pegIFN alpha-2a 180 mcg subcutaneously once weekly and RBV 1000 mg/day if participant weighed <=75 kg or RBV 1200 mg/day if participant weighed > 75 kg, orally in 2 divided doses up to Week 48 and then followed through Week 72.
- Placebo Plus pegIFN/RBV: Placebo matched to filibuvir tablet orally twice daily as blinded therapy in combination with pegIFN alpha-2a 180 mcg subcutaneously once weekly and RBV 1000 mg/day to participants weighing <=75 kg or RBV 1200 mg/day to participants weighing >75 kg, orally in 2 divided doses up to Week 24 followed by open-label pegIFN alpha-2a 180 mcg subcutaneously once weekly and RBV 1000 mg/day to participants weighing <=75 kg or RBV 1200 mg/day to participants weighing >75 kg orally in 2 divided doses up to Week 48. Participants were then followed through Week 72.
Period: Overall Study
Arm/Group | Filibuvir 300 mg Plus pegIFN/RBV | Filibuvir 600 mg Plus pegIFN/RBV | Placebo Plus pegIFN/RBV
Started | 96 | 96 | 96
Completed | 39 | 41 | 45
Not Completed | 57 | 55 | 51
Not completed — Adverse Event | 10 | 9 | 8
Not completed — Insufficient Virologic Response | 10 | 7 | 12
Not completed — Virologic Breakthrough | 2 | 2 | 8
Not completed — Lost to Follow-up | 10 | 6 | 2
Not completed — Withdrawal by Subject | 6 | 9 | 9
Not completed — Other | 0 | 2 | 5
Not completed — Protocol Violation | 1 | 0 | 2
Not completed — Participant Relapsed | 18 | 20 | 5

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all randomized participants who took at least 1 dose of study drug.
Groups:
- Filibuvir 300 mg Plus pegIFN/RBV: Filibuvir 300 mg tablet orally twice daily as blinded therapy along with pegIFN alpha-2a 180 mcg subcutaneously once weekly and RBV 1000 mg/day to participants weighing <=75 kg or RBV 1200 mg/day to participants weighing >75 kg orally in 2 divided doses up to Week 24. Participants with undetectable HCV RNA (plasma HCV RNA <15 IU/mL) from Week 4 through 24 were discontinued from therapy and followed through Week 72. Participants with detectable HCV RNA (>=15 IU/mL) at Week 4 or later but undetectable at Week 24 received open-label pegIFN alpha-2a 180 mcg subcutaneously once weekly and RBV 1000 mg/day if participant weighed <=75 kg or RBV 1200 mg/day if participant weighed > 75 kg, orally in 2 divided doses up to Week 48 and then followed through Week 72.
- Total: Total of all reporting groups
Arm/Group | Filibuvir 300 mg Plus pegIFN/RBV | Filibuvir 600 mg Plus pegIFN/RBV | Placebo Plus pegIFN/RBV | Total
Number analyzed (Participants) | 96 | 96 | 96 | 288
Age, Customized [Number; unit: participants]
  18 to 44 years | 36 | 25 | 31 | 92
  45 to 64 years | 56 | 68 | 61 | 185
  >=65 years | 4 | 3 | 4 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 47 | 44 | 135
  Male | 52 | 49 | 52 | 153

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Viral Response (SVR) at Week 72
Description: For participants who received filibuvir, had undetectable HCV RNA from Week 4 through 24 and discontinued therapy at Week 24, SVR was defined as undetectable plasma HCV RNA levels (<15 IU/mL) at both Week 24 (End of Treatment [EOT]) and Week 72, regardless of the HCV RNA levels between Week 24 and 72. For participants who received filibuvir, had detectable HCV RNA at Week 4 or later and discontinued therapy at Week 48 or who received placebo, SVR was defined as undetectable plasma HCV RNA levels (<15 IU/mL) at both Week 48 (EOT) and Week 72, regardless of the HCV RNA levels between Week 48 and 72.
Time Frame: Week 72
Population: ITT population included all randomized participants who took at least 1 dose of study drug. If a participant had a missing value at Week 72, participant was considered a failure; if a participant had achieved SVR but died or discontinued within same time period, the participant was considered a success.
Measure: Number; unit: percentage of participants
Arm/Group | Filibuvir 300 mg Plus pegIFN/RBV | Filibuvir 600 mg Plus pegIFN/RBV | Placebo Plus pegIFN/RBV
Number analyzed (Participants) | 96 | 96 | 96
percentage of participants | 41.7 | 39.6 | 45.8

2. Secondary Outcome: Percentage of Participants With Undetectable Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) at Week 4, 12, 24 and 48
Description: Percentage of participants with undetectable HCV RNA at Week 4 (rapid viral response [RVR]), Week 12 (early viral response [EVR]), Week 24 and Week 48 were summarized. Undetectable HCV RNA was defined as plasma HCV RNA levels <15 IU/mL.
Time Frame: Week 4, 12, 24, 48
Population: ITT population included all randomized participants who took at least 1 dose of study drug. Last observation carried forward (LOCF) method was used to impute missing values for participants who did not discontinue from study. Participants who discontinued early from the study were considered not to have undetectable HCV RNA.
Measure: Number; unit: percentage of participants
Arm/Group | Filibuvir 300 mg Plus pegIFN/RBV | Filibuvir 600 mg Plus pegIFN/RBV | Placebo Plus pegIFN/RBV
Number analyzed (Participants) | 96 | 96 | 96
percentage of participants
  Week 4 | 58.3 | 61.5 | 28.1
  Week 12 | 76.0 | 78.1 | 67.7
  Week 24 | 74.0 | 76.0 | 77.1
  Week 48 | 54.2 | 58.3 | 64.6

3. Secondary Outcome: Percentage of Participants With Sustained Viral Response at 12 Weeks Following Completion of Therapy (SVR12)
Description: A participant was considered to have achieved SVR12 if the plasma HCV RNA levels were <15 IU/mL at both the end of treatment (Week 24 or 48, depending on the time of therapy discontinuation based on HCV RNA levels during therapy) and 12 weeks following the completion of therapy (Week 36 for participants who ended therapy at Week 24; Week 60 for participants who ended therapy at Week 48). Overall percentage of participants with SVR12 was summarized.
Time Frame: 12 weeks after completion of therapy (Week 36 or 60)
Population: ITT population. Participant with missing HCV RNA values at end of treatment and all follow-up visits or at the specified time point and all subsequent visits was considered not to have undetectable HCV RNA. Missing HCV RNA value at 12 weeks following completion of therapy was imputed using value of subsequent follow-up visit, if available.
Measure: Number; unit: percentage of participants
Arm/Group | Filibuvir 300 mg Plus pegIFN/RBV | Filibuvir 600 mg Plus pegIFN/RBV | Placebo Plus pegIFN/RBV
Number analyzed (Participants) | 96 | 96 | 96
percentage of participants | 42.7 | 44.8 | 45.8

4. Secondary Outcome: Percentage of Participants With Sustained Viral Response at 24 Weeks Following Completion of Therapy (SVR24)
Description: SVR24 was summarized only for those participants who received filibuvir, had undetectable HCV RNA from Week 4 through 24 and discontinued therapy at Week 24 and all participants who received placebo for 48 weeks. A participant was considered to have achieved SVR24 if the plasma HCV RNA levels were <15 IU/mL at both the end of treatment (Week 24 for filibuvir participants who ended therapy at Week 24 and Week 48 for participants who received placebo) and 24 weeks following the completion of therapy (Week 48 for filibuvir participants who ended therapy at Week 24; Week 72 for placebo participants who ended therapy at Week 48).
Time Frame: 24 weeks after completion of therapy (Week 48 or 72)
Population: ITT population.N (number of participants analyzed)=evaluable participants for the measure. Missing HCV RNA value at EOT, all follow-up visits/at specified time point, all subsequent visits was considered not to have undetectable HCV RNA.Missing HCV RNA value at 24 weeks after EOT was imputed using value of subsequent follow-up visit, if available.
Measure: Number; unit: percentage of participants
Groups:
- Filibuvir 300 mg Plus pegIFN/RBV: Filibuvir 300 mg tablet orally twice daily as blinded therapy along with pegIFN alpha-2a 180 mcg subcutaneously once weekly and RBV 1000 mg/day to participants weighing <=75 kg or RBV 1200 mg/day to participants weighing >75 kg orally in 2 divided doses up to Week 24. Participants with undetectable HCV RNA (plasma HCV RNA <15 IU/mL) from Week 4 through 24 were discontinued from therapy and followed through Week 72.
- Filibuvir 600 mg Plus pegIFN/RBV: Filibuvir 600 mg tablet orally twice daily as blinded therapy along with pegIFN alpha-2a 180 mcg subcutaneously once weekly and RBV 1000 mg/day to participants weighing <=75 kg or RBV 1200 mg/day to participants weighing >75 kg orally in 2 divided doses up to Week 24. Participants with undetectable HCV RNA (plasma HCV RNA <15 IU/mL) from Week 4 through 24 were discontinued from therapy and followed through Week 72.
Arm/Group | Filibuvir 300 mg Plus pegIFN/RBV | Filibuvir 600 mg Plus pegIFN/RBV | Placebo Plus pegIFN/RBV
Number analyzed (Participants) | 45 | 47 | 67
percentage of participants | 73.3 | 66.0 | 65.7

5. Secondary Outcome: Percentage of Participants With Breakthrough Viremia
Description: A participant was considered to have breakthrough viremia if there was a >2 log10 increase from nadir in HCV RNA concentration while on treatment or HCV RNA that became undetectable with treatment but then became persistently detectable (2 or more consecutive viral RNA measurements >1000 IU/mL) again during treatment. Overall percentage of participants with breakthrough viremia was summarized.
Time Frame: Baseline up to Week 48
Population: ITT population included all randomized participants who took at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Filibuvir 300 mg Plus pegIFN/RBV | Filibuvir 600 mg Plus pegIFN/RBV | Placebo Plus pegIFN/RBV
Number analyzed (Participants) | 96 | 96 | 96
percentage of participants | 4.2 | 4.2 | 7.3

6. Secondary Outcome: Percentage of Participants With Relapsed Response
Description: A participant was considered to have relapsed response if the plasma HCV RNA levels were undetectable at end of treatment (Week 24 or 48, depending on the time of therapy discontinuation based on HCV RNA levels during therapy) but detectable (>=15 IU/mL) during the off-treatment follow-up period up to Week 72. Overall percentage of participants with relapsed response was summarized.
Time Frame: Week 24 or Week 48 up to Week 72
Population: ITT population included all randomized participants who took at least 1 dose of study drug. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. Participant with all the HCV RNA values missing during follow-up was imputed as having relapsed.
Measure: Number; unit: percentage of participants
Arm/Group | Filibuvir 300 mg Plus pegIFN/RBV | Filibuvir 600 mg Plus pegIFN/RBV | Placebo Plus pegIFN/RBV
Number analyzed (Participants) | 64 | 70 | 59
percentage of participants | 35.9 | 42.9 | 25.4

7. Secondary Outcome: Change From Baseline in Plasma Log10 Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) at Week 4, 12 and 24
Description: Plasma HCV RNA levels were measured using the Roche COBAS TaqMan assay (limit of detection: 15 IU/mL). Baseline value calculated as the average of the screening and Day 1 pre-dose measurements.
Time Frame: Baseline, Week 4, 12, 24
Population: ITT population included all randomized participants who took at least 1 dose of study drug. LOCF method was used for imputing missing values for participants who did not discontinue from study. Final value was imputed as baseline for participants who discontinued before the time point of interest.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Filibuvir 300 mg Plus pegIFN/RBV | Filibuvir 600 mg Plus pegIFN/RBV | Placebo Plus pegIFN/RBV
Number analyzed (Participants) | 96 | 96 | 96
log10 IU/mL
  Baseline | 6.1 (0.7) | 6.0 (0.6) | 6.1 (0.7)
  Change at Week 4 | -4.0 (1.6) | -4.2 (1.2) | -3.0 (1.6)
  Change at Week 12 | -4.1 (1.8) | -4.2 (1.6) | -3.9 (1.7)
  Change at Week 24 | -3.7 (2.2) | -3.8 (2.1) | -3.9 (2.0)

8. Secondary Outcome: Number of Adverse Events (AEs) by Severity (All Causality)
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. A serious AE (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Adverse events were graded as mild (did not interfere with participant's usual function), moderate (interfered to some extent with participant's usual function) or severe (interfered significantly with participant's usual function). The most severe grade was used in case of multiple occurrences of the same event.
Time Frame: Baseline up to Week 72
Population: Safety population included all randomized participants who took at least 1 dose of study drug analyzed as treated.
Measure: Number; unit: adverse events
Arm/Group | Filibuvir 300 mg Plus pegIFN/RBV | Filibuvir 600 mg Plus pegIFN/RBV | Placebo Plus pegIFN/RBV
Number analyzed (Participants) | 96 | 96 | 96
adverse events
  Mild | 672 | 731 | 745
  Moderate | 154 | 169 | 179
  Severe | 35 | 20 | 27

9. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) by Relationship to Study Drug (Any Therapy)
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to Week 72 that were absent before treatment or that worsened relative to pretreatment state. All causality AEs included SAEs as well as non-serious AEs, without regard to relationship to the study drug, which occurred during the trial. Treatment-related were events considered related to study drug by the investigator. Number of participants with treatment related TEAEs and all causality TEAEs were summarized.
Time Frame: Baseline up to Week 72
Population: Safety population included all randomized participants who took at least 1 dose of study drug analyzed as treated.
Measure: Number; unit: participants
Arm/Group | Filibuvir 300 mg Plus pegIFN/RBV | Filibuvir 600 mg Plus pegIFN/RBV | Placebo Plus pegIFN/RBV
Number analyzed (Participants) | 96 | 96 | 96
participants
  Treatment related AEs | 85 | 88 | 91
  All-causality AEs | 88 | 92 | 92

10. Secondary Outcome: Number of Participants Who Discontinued Study Due to Adverse Events (AEs)
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Baseline up to Week 72
Population: Safety population included all randomized participants who took at least 1 dose of study drug analyzed as treated.
Measure: Number; unit: participants
Arm/Group | Filibuvir 300 mg Plus pegIFN/RBV | Filibuvir 600 mg Plus pegIFN/RBV | Placebo Plus pegIFN/RBV
Number analyzed (Participants) | 96 | 96 | 96
participants | 10 | 9 | 8

11. Secondary Outcome: Number of Participants With Dose Reduction or Temporary Discontinuation Due to Adverse Events (AEs)
Description: as for outcome 10
Time Frame: Baseline up to Week 72
Population: Safety population included all randomized participants who took at least 1 dose of study drug analyzed as treated.
Measure: Number; unit: participants
Arm/Group | Filibuvir 300 mg Plus pegIFN/RBV | Filibuvir 600 mg Plus pegIFN/RBV | Placebo Plus pegIFN/RBV
Number analyzed (Participants) | 96 | 96 | 96
participants | 28 | 22 | 28

12. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities by Severity
Description: Number of participants with laboratory abnormalities by Division of Auto Immune Disease Syndrome (DAIDS) grade of 4; 3 or 4; 2, 3 or 4 was summarized. Abnormal laboratory values refers to a DAIDS grade greater than 0, where grade 1= mild, grade 2= moderate, grade 3= severe and grade 4 = potentially life-threatening.
Time Frame: Baseline up to Week 72
Population: Safety population included all randomized participants who took at least 1 dose of study drug analyzed as treated. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Filibuvir 300 mg Plus pegIFN/RBV | Filibuvir 600 mg Plus pegIFN/RBV | Placebo Plus pegIFN/RBV
Number analyzed (Participants) | 94 | 96 | 96
participants
  Grade 4 | 11 | 16 | 8
  Grade 3 or 4 | 37 | 46 | 43
  Grade 2, 3 or 4 | 73 | 83 | 81

13. Secondary Outcome: Plasma Concentration of Filibuvir, Pegylated Interferon and Ribavirin
Time Frame: Week 0 (pre-dose), Week 2, 4, 8, 12, 16, 20, 24, 48 (only for those participants who received treatment till Week 48) post-dose
Population: Data could not be summarized due to sparse sampling time points adopted for this study.
Arm/Group | Filibuvir 300 mg Plus pegIFN/RBV | Filibuvir 600 mg Plus pegIFN/RBV | Placebo Plus pegIFN/RBV
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Filibuvir 300 mg Plus pegIFN/RBV | Filibuvir 600 mg Plus pegIFN/RBV | Placebo Plus pegIFN/RBV
Serious Adverse Events (participants affected / at risk) | 14/96 | 6/96 | 6/96
Other Adverse Events (participants affected / at risk) | 85/96 | 89/96 | 90/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Filibuvir 300 mg Plus pegIFN/RBV (N=96) | Filibuvir 600 mg Plus pegIFN/RBV (N=96) | Placebo Plus pegIFN/RBV (N=96)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Vestibular disorder (Ear and labyrinth disorders) | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 1
Bacterial abscess central nervous system (Infections and infestations) | 0 | 1 | 0
Lymph node tuberculosis (Infections and infestations) | 1 | 0 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Actinomyces test positive (Investigations) | 0 | 1 | 0
Blood urea nitrogen/creatinine ratio increased (Investigations) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Cardiac neurosis (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary calcification (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Filibuvir 300 mg Plus pegIFN/RBV (N=96) | Filibuvir 600 mg Plus pegIFN/RBV (N=96) | Placebo Plus pegIFN/RBV (N=96)
Anaemia (Blood and lymphatic system disorders) | 15 | 11 | 16
Leukopenia (Blood and lymphatic system disorders) | 4 | 5 | 6
Lymphopenia (Blood and lymphatic system disorders) | 5 | 3 | 3
Neutropenia (Blood and lymphatic system disorders) | 15 | 11 | 20
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 6 | 3
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 5
Vertigo (Ear and labyrinth disorders) | 2 | 3 | 5
Hypothyroidism (Endocrine disorders) | 0 | 2 | 6
Dry eye (Eye disorders) | 2 | 3 | 5
Vision blurred (Eye disorders) | 3 | 5 | 5
Abdominal pain (Gastrointestinal disorders) | 6 | 3 | 4
Abdominal pain upper (Gastrointestinal disorders) | 11 | 10 | 4
Aphthous stomatitis (Gastrointestinal disorders) | 2 | 7 | 4
Constipation (Gastrointestinal disorders) | 7 | 3 | 10
Diarrhoea (Gastrointestinal disorders) | 14 | 10 | 17
Dry mouth (Gastrointestinal disorders) | 7 | 7 | 4
Dyspepsia (Gastrointestinal disorders) | 5 | 6 | 7
Nausea (Gastrointestinal disorders) | 20 | 35 | 30
Stomatitis (Gastrointestinal disorders) | 3 | 2 | 5
Vomiting (Gastrointestinal disorders) | 9 | 11 | 13
Asthenia (General disorders) | 16 | 19 | 20
Chills (General disorders) | 11 | 14 | 12
Fatigue (General disorders) | 36 | 37 | 36
Influenza like illness (General disorders) | 15 | 14 | 19
Injection site reaction (General disorders) | 4 | 4 | 5
Irritability (General disorders) | 14 | 19 | 15
Oedema peripheral (General disorders) | 2 | 7 | 4
Pain (General disorders) | 4 | 5 | 8
Pyrexia (General disorders) | 14 | 14 | 15
Bronchitis (Infections and infestations) | 4 | 5 | 1
Influenza (Infections and infestations) | 3 | 4 | 5
Weight decreased (Investigations) | 13 | 7 | 5
White blood cell count decreased (Investigations) | 0 | 1 | 5
Decreased appetite (Metabolism and nutrition disorders) | 20 | 16 | 23
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 17 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 8 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 17 | 20 | 25
Disturbance in attention (Nervous system disorders) | 2 | 7 | 1
Dizziness (Nervous system disorders) | 12 | 8 | 12
Dysgeusia (Nervous system disorders) | 16 | 24 | 5
Headache (Nervous system disorders) | 28 | 33 | 35
Syncope (Nervous system disorders) | 5 | 1 | 1
Anxiety (Psychiatric disorders) | 6 | 3 | 7
Depression (Psychiatric disorders) | 21 | 10 | 12
Insomnia (Psychiatric disorders) | 24 | 31 | 28
Sleep disorder (Psychiatric disorders) | 5 | 2 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 18 | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 9 | 18
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 18 | 16 | 24
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 20 | 13 | 19
Eczema (Skin and subcutaneous tissue disorders) | 6 | 5 | 2
Erythema (Skin and subcutaneous tissue disorders) | 3 | 5 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 1 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 27 | 29 | 19
Rash (Skin and subcutaneous tissue disorders) | 12 | 22 | 18
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.